CLINICAL TRIAL: NCT02620592
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ZYDPLA1, a Novel DPP- IV Inhibitor, Following Oral Administration in Healthy Volunteers
Brief Title: Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics (PKs) of ZYDPLA1 Following Oral Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: ZYDPLA1 1001
Record Dates: First submitted 2015-11-24; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes Mellitus
Keywords: Healthy Subject; ZYDPLA1; DPPIV inhibitor; Pharmacokinetics; Safety
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZYDPLA1 tablet (Active Comparator): ZYDPLA1 tablets: Route of administration: Oral Dosage (Single Ascending Study): 1 mg, 5mg, 20mg, 50mg, 100mg, 200mg Multiple Ascending Study: 100mg, 200mg Food effect and Gender effect study: 200mg
  Interventions: Drug: ZYDPLA1 tablet
- Placebo (Placebo Comparator): Placebo tablets: Route of administration: Oral Dosage (Single Ascending Study): 1 mg, 5mg, 20mg, 50mg, 100mg, 200mg Multiple Ascending Study: 100mg, 200mg Food effect and Gender effect study: 200mg
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: ZYDPLA1 tablet — The oral dose of ZYDPLA1 tablet administered with 240 ± 10 mL of water at ambient temperature.
  Arms: ZYDPLA1 tablet
Drug: Placebo tablet — The oral dose of placebo tablet administered with 240 ± 10 mL of water at ambient temperature.
  Arms: Placebo

SUMMARY:
This First in Human (FIH) Phase I study intends to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of ZYDPLA1 in normal healthy adult volunteers.

DETAILED DESCRIPTION:
Glucose-dependent insulinotropic polypeptide (GIP) and Glucagon-like peptide (GLP-1) are incretin hormones, which stimulate glucose dependent insulin secretion, inhibit glucagon secretion, delay gastric emptying, suppress appetite and improve peripheral glucose uptake and disposal. Dipeptidyl peptidase-IV (DPP-IV) is a serine protease, which selectively cleaves the first two amino acids of GIP and GLP-1 thereby making it inactive. Inhibition of DPP-IV activity elevates endogenous GIP, GLP-1 and insulin levels thereby improving glucose excursion and exhibits antidiabetic activity. Since no orally active GLP-1 agonists are available, clinically orally bioavailable DPP-IV inhibitors hold great potential for the treatment of type 2 diabetes mellitus.

Cadila Healthcare Ltd. developed a novel and orally bioavailable DPP-IV inhibitor (ZYDPLA1). In-vitro studies confirm selective DPPIV inhibitory activity of the ZYDPLA1. Pre-clinical in vivo pharmacodynamic, absorption, distribution, metabolism and excretion (ADME) & toxicological studies showed the promising antidiabetic activity, good exposure and safety profile of ZYDPLA1(in various animal models).

Hence a randomized, double-blind, placebo-controlled first in man trial proposed to evaluate the safety and tolerability of ZYDPLA1 in healthy volunteers.

This study included 4 plans:

i) single dose escalation study ii) multiple dose escalation study, iii) gender effect study and iv) food effect study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female between 18 and 65 years of age.
2. Male subjects must agree to use one of the contraception methods during the study. Male contraceptive options include: Vasectomy, Abstinence requiring the use of contraceptives if becoming sexually active, or double barrier method (condom with spermicide, diaphragm or cervical cap). No Sperm donation for at least up to 90 days after last investigational product.
3. BMI within the range 18.0 - 30.0 kg/m2 BMI value should be rounded off to one significant digit after decimal point. BMI values should be rounded to the nearest integer (ex. 30.4 rounds down to 30, while 17.5 rounds up to 18).
4. Capable of giving written informed consent, which includes compliance with protocol.
5. Corrected QT interval (QTc) interval < 450msec (as measured by QTcF)
6. For gender effect study, only females with history of sterility or at least 1 year menopause or use of long acting non hormonal contraceptive measures (e.g., intrauterine device) will be recruited. Surgical sterility is defined as either bilateral tubal ligation/occlusion, bilateral oophorectomy or hysterectomy.
7. Negative Urine drug screen including amphetamine, barbiturates, benzodiazepines, cannabinoid, cocaine, opiates, methadone and phencyclidine within 28 days prior to initiation of the study and prior to check-in.

Exclusion Criteria:

1. Presence or history of pancreatitis at any time {Serum Amylase/Serum Lipase more than significant upper normal limit (≥1.5 times UNL)}
2. Presence or history of severe gastrointestinal disease in the last 6 months
3. Presence or history of renal insufficiency at any time {Serum creatinine more than upper normal limit (UNL)}
4. Active liver disease and/or liver transaminases greater than 1.5 times UNL
5. History or presence of other systemic disorders or diseases (e.g., respiratory, gastrointestinal, endocrine, immunological, dermatological, neurological, psychiatric disease or any other body system involvement)
6. History or presence of any medication in the last 14 days
7. History or presence of significant alcoholism or drug abuse within the past 1 year
8. History or presence of significant smoking (more than 10 cigarettes per day) or consumption of tobacco products (more than 10 times per day)
9. Difficulty with donating blood or difficulty in accessibility of veins.
10. Intolerance to venipuncture.
11. Systolic blood pressure more than 150 mmHg and less than 100 mmHg and diastolic blood pressure more than 90 mmHg
12. Pulse rate less than 50/minute and more than 100/minute
13. Any clinically significant laboratory findings during screening
14. History or presence of any clinically significant electrocardiogram (ECG) abnormalities during screening as determined by the Principal Investigator.
15. Major illness and/or major surgery in last 3 months
16. Volunteers who have participated in any drug research study other than the present trial within the past 30 days (Subjected to Insurance that subject has not participated in long acting drug including new biological entities/new chemical entities/biosimilar products).
17. Volunteers who have donated one unit (450 mL) of blood in the past 3 months
18. Positive Alcohol breath analyzer at the time of Screening and Check-in
19. A positive hepatitis screen (includes subtype B and C) and/or a positive test result for HIV antibody.
20. Any food allergy, intolerance, restriction or special diet that, in the opinion of the Principal investigator or Sub-investigator, could contraindicate the study participant's participation in this study.
21. For gender effect study, female volunteers with following criteria will not be recruited:

    * History of pregnancy or lactation in the past 3 months
    * Fertile female volunteers not protected against pregnancy by adequate long-term anti-fertility measures
    * History of less than 1 year of menopause and not using adequate long-term antifertility measures
    * Using hormonal contraceptives
    * Using hormone replacement therapy
    * Unable to give assurance for protection against pregnancy for 3 months after the participation in this trial
    * Positive urine pregnancy test on the day of check-in (women of child bearing potential)
    * Positive serum β-human chorionic gonadotropin (hCG) level at the screening visit (women of child bearing potential)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by monitoring adverse events, clinical, laboratory, electrocardiogram, and vital signs examinations. | 14 Days (Plan 1, III, and IV);
Safety and tolerability assessed by monitoring adverse events, clinical, laboratory, electrocardiogram, and vital signs examinations. | 28 Days (Plan II)

SECONDARY OUTCOMES:
Pharmacokinetic assessment: Maximum plasma concentration (Cmax) | 14 Days (Plan I, III, and IV)
Maximum plasma concentration (Cmax) | 28 Days (Plan II)
Time to reach maximum plasma concentration (Tmax) | 14 Days (Plan I, III, and IV)
Time to reach maximum plasma concentration (Tmax) | 28 Days (Plan II)
Area under the curve from the time of dosing to the last measurable concentration (AUC0-t) | 14 Days (Plan I, III, and IV)
Area under the curve from the time of dosing to the last measurable concentration (AUC0-t) | 28 Days (Plan II)
Area under the curve from the time of dosing to the infinity (AUC 0-inf) | 14 Days (Plan I, III, and IV)
Area under the curve from the time of dosing to the infinity (AUC 0-inf) | 28 Days (Plan II)
Terminal half life (t1/2) | 14 Days (Plan I, III, and IV)
Terminal half life (t1/2) | 28 Days (Plan II)
Elimination rate constant (λz) | 14 Days (Plan I, III, and IV)
Elimination rate constant (λz) | 28 Days (Plan II)
Clearance (CL) | 14 Days (Plan I, III, and IV)
Clearance (CL) | 28 Days (Plan II)
Volume of distribution (Vd) | 14 Days (Plan I, III, and IV)
Volume of distribution (Vd) | 28 Days (Plan II)
Accumulation index | 28 Days (Plan II)
Pharmacodynamic effect (Plan I, III, and IV) assessment by monitoring primary parameters: Plasma DPPIV | 14 Days
Pharmacodynamic effect (Plan II) assessment by monitoring primary parameters: Plasma DPPIV | 28 Days
Glucagon-like peptide-1 (active and total) | 14 Days
Glucagon-like peptide-1 (active and total) | 28 Days
Secondary parameters: Plasma glucose | 14 Days
Plasma glucose | 28 Days
Serum insulin | 14 Days
Serum insulin | 28 Days
C-peptide | 14 Days
C-peptide | 28 Days
Glucagon | 14 Days
Glucagon | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Rajendrakumar H Jani, Ph.D.,, Study Director — Zydus Lifesciences Limited
Locations (1):
- Profil Institute for Clinical Research, Chula Vista, California, United States